CLINICAL TRIAL: NCT00715494
Title: Returning to Everyday Tasks Utilizing Rehabilitation Networks (RETURN)
Brief Title: A Pilot Study of Rehabilitation Among Intensive Care Unit (ICU) Survivors: the RETURN Trial
Acronym: RETURN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University School of Medicine (Other); Duke University (Other); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wes Ely, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 070971
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Brain Injury; Muscle Weakness
Keywords: brain injuries, dementia, myopathies, muscle disorders
MeSH Terms: conditions — Brain Injuries; Muscle Weakness; Dementia; Muscular Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: This was a single-site, feasibility, pilot, randomized trial of 21 general medical/surgical intensive care unit survivors (8 controls and 13 intervention patients) with either cognitive or functional impairment at hospital discharge. After discharge, study controls received usual care (sporadic rehabilitation), whereas intervention patients received a combination of in-home cognitive, physical, and functional rehabilitation over a 3-month period via a social worker or master's level psychology technician utilizing telemedicine to allow specialized multidisciplinary treatment. Interventions over 12 wks included six in-person visits for cognitive rehabilitation and six televisits for physical/functional rehabilitation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Control (No Intervention): Patients (Controls) will not receive formal (study-related) rehabilitation interventions and will only receive usual care.
- Group 2 - Intervention (Experimental): Participants in the experimental group will receive a focused set of interdisciplinary home-based interventions over a 12 week period.
  Interventions: Behavioral: Cognitive, physical, and functional rehabilitation

INTERVENTIONS:
Behavioral: Cognitive, physical, and functional rehabilitation — A multicomponent program of cognitive, physical, and functional rehabilitation interventions will be delivered to patients in their home environments over a focused 12 week period with the aid of tele-technology to utilize the expertise of physical therapy, occupational therapy, and neuropsychology.
  Arms: Group 2 - Intervention

SUMMARY:
Intensive care unit (ICU) hospitalization saves lives but often does so at a high personal cost to ICU survivors who frequently experience significant cognitive impairment and an array of physical and functional disabilities that limit their recovery and quality of life. While the problems experienced by these patients are likely amenable to rehabilitation, few ICU survivors receive focused rehabilitation following hospital discharge. The purpose of this study is to initiate and test the feasibility of a complex intervention incorporating a cognitive, physical, and functional rehabilitation program at the time of hospital discharge and implement this 12 week program using in-home visits and tele-technology. We hypothesize that this interdisciplinary rehabilitation program, initiated at hospital discharge and implemented using in-home visits and tele-technology, will result in improved recovery of neuropsychological and physical performance and overall functional status.

DETAILED DESCRIPTION:
The long-term consequences of critical illness and intensive care unit (ICU) hospitalization in ICU survivors are profound and include cognitive, physical, and functional impairments. The purpose of this study is to pilot test a 12-week, home-based rehabilitation program targeting both cognitive functioning and physical functioning, to determine the feasibility of such a rehabilitation program, and to determine whether participation in a rehabilitation program will result in improved outcomes among ICU survivors. The study will rely on a randomized controlled clinical trial design, with patients assigned to either a "usual care" control group vs. the treatment group. Individuals in the treatment group will receive a protocolized cognitive rehabilitation intervention, as well as individualized physical and functional rehabilitation targeted at abilities such as strength, endurance, balance, and functionality in basic tasks of daily living. Cognitive, physical, and functional rehabilitation interventions will be delivered in patient homes and will take place on alternating weeks over a 12 week period. Televideo technology will be employed in the context of these interventions, with experts from Vanderbilt University and Duke University medical centers providing assistance via a video monitor in conjunction with a rehabilitation specialist who will implement interventions in patient homes. The study has 3 primary outcomes including: (1). Executive functioning (e.g. ability to plan, organize, multi-task) over time as measured by the Tower Test, a psychometric tool evaluating executive abilities; (2) Physical Impairment, as measured by the Timed Up and Go (TUG) test; (3) Physical Functioning, as measured by the Step Activity Monitor (SAM). These three primary outcomes have been selected as areas of primary focus due to the fact that available research points to the presence of significant deficits in these areas among ICU survivors. Secondary outcomes include activities of daily living (Katz ADL) and instrumental activities of daily living (Pfeffers FAQ), activity specific balance and confidence(ABC Scale), health related quality of life (SF-36), 12-month mortality, and both rehospitalization rates and number of rehospitalization days. We will measure change in the outcome measures of interest at 3 and 12-month follow up to determine short term efficacy, along with evaluating overall feasibility. The study duration will include 1 year of protocol development for the complex intervention and 1.5 to 2 years of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the BRAIN-ICU study (AG027472-01A1), the presence of cognitive impairment defined via an abnormal Tower Test score (at the time of hospital discharge) and/or physical impairment defined per standard cutpoints for the Timed Up and Go Test (at the time of hospital discharge);
* The ability to walk with or without assistance.

Exclusion Criteria:

* Moderate to severe dementia on ICU admission based on a standardized surrogate assessment (as this would prohibit patients from functioning independently at home);
* The presence of normal cognition and normal physical function at the time of screening (i.e. hospital discharge) which would eliminate the need for rehabilitation;
* Lacking telephone service with an analog telephone line (which would preclude the tele-video component of the RETURN intervention).
* Live greater than 125 miles from Nashville
* Patient is unable to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tower Test - a psychometric measure of executive functioning | 3 and 12 months post hospital discharge
Timed Up and Go (TUG), a timed test assessing physical strength and gait speed | 3 and 12 months post-hospital discharge
Step Activity Monitor (SAM), a device that measures total level of participant activity | 3 and 12 months post-hospital discharge

SECONDARY OUTCOMES:
Pfeffers FAQ, a brief measure of higher order (IADL) functioning. | 3 and 12 months post-hospital discharge
SF-36 global scores | 3 and 12 months post hospital discharge
Katz Activities of Daily Living (ADL) scale | 3 and 12 months post hospital discharge
Activities-specific Balance Confidence Scale (ABC) | 3 and 12 months post hospital discharge
Mortality | Within 12 months of hospital discharge
Rehospitalization rate and number of hospital days | Within 12 months of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: E Wesley Ely, MD, MPH, Principal Investigator — Vanderbilt University School of Medicine; Helen Hoenig, MD, MPH, Principal Investigator — Duke University Medical Center, Durham VA Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- See also: ICU Delirium and Cognitive Impairment Study Group — http://www.icudelirium.org